CLINICAL TRIAL: NCT01731119
Title: An Open-Label Pilot Study of Lurasidone in Treating Antipsychotic Naive or Quasi-Naive Children and Adolescents
Brief Title: Study of Lurasidone in Treating Antipsychotic Naive or Quasi-Naive Children and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-2302
Record Dates: First submitted 2012-11-14; First posted 2012-11-21 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Psychosis NOS; Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive; Bipolar I Disorder; Bipolar II Disorder; Mood Disorder NOS; Severe Major Depression With Psychotic Features; Single Episode Major Depression Without Psychotic Symptoms; Severe Mood Disorder With Psychotic Features
Keywords: Latuda,lurasidone,antipsychotics,autism, mood, psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders; Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive; Bipolar Disorder; Mood Disorders | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flexible Dose Latuda© (Experimental): Lurasidone (Latuda©)dose will be determined solely by the clinician in accordance with the best interests of each participant.
  Interventions: Drug: Latuda©

INTERVENTIONS:
Drug: Latuda© — All subjects will be started on 20-40mg of Latuda© at night (suggested intake with food). Subsequently, the dose may be increased as clinically indicated and based on tolerability every 7 days by 20-40mg to a maximum of 160mg per day with food which may be given as a single or twice daily dose depending on participant's preference. The maintenance dose will be determined solely by the clinician in accordance with the best interests of each participant.
  Other Names: Lurasidone Hydrochloride tablets

SUMMARY:
The overarching purpose of this pilot study is to collect preliminary data regarding the variability of weight gain associated with lurasidone (Latuda©) treatment of antipsychotic naive children and adolescents in order to inform decisions about including a lurasidone arm in a future large scale trial of different approaches to minimize antipsychotic associated weight gain in the pediatric population. In adults, lurasidone appears to cause minimal weight gain. The participants will be 6-19 years old with psychotic spectrum, mood spectrum, or autism spectrum disorders. They will have 4 weeks or less of lifetime antipsychotic exposure.

DETAILED DESCRIPTION:
This is a multi-site, 12-week, open-label study assessing the weight and metabolic changes associated with lurasidone treatment. Antipsychotic (AP) naive subjects will start open-label treatment by following a flexible titration schedule. Quasi-antipsychotic naive subjects (less than 4 weeks of total AP treatment) will be started on lurasidone and tapered off the other antipsychotic over an estimated 4 weeks depending on the dose and tolerability of the prior antipsychotic. Other psychoactive medications including antidepressants, benzodiazepines, stimulants, alpha-2 agonists, and mood stabilizers are allowed as long as the dose is not changed, unless it is clinically necessary. Assessments of weight, efficacy, and side effects are conducted at baseline, week 2, week 4, week 8, and week 12. The primary outcome is percent change in weight. The secondary outcomes include psychiatric efficacy measures and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children and adolescents between 6 and 19 years of age of any race or ethnicity
* Subject must meet Diagnostic Statistical Manual (DSM)-IV-Text Revision (TR) criteria for a psychotic spectrum, mood spectrum or autism spectrum disorder as defined by one of the following diagnoses:

  * schizophrenia (any type)
  * schizoaffective disorder
  * schizophreniform disorder
  * psychosis Not Otherwise Specified (NOS)
  * autistic disorder with significant irritability/aggression (Aberrant Behavioral Checklist-Community (ABC-C) Irritability subscale score of greater than or equal to 18)
  * Asperger syndrome with significant irritability/aggression (ABC-C Irritability subscale score of greater than or equal to 18)
  * pervasive developmental disorder NOS with significant irritability/aggression (ABC-C Irritability subscale score of greater than or equal to 18)
  * bipolar type I
  * bipolar type II
  * mood disorder NOS
  * major depression with psychotic features
  * major depression (unresponsive to 2 different antidepressants)
  * severe mood dysregulation (SMD) according to Leibenluft and colleagues broad spectrum bipolar disorder
* Subjects must have ≤ 4 weeks of lifetime exposure to an antipsychotic medication at any dosage. These medications include olanzapine (Zyprexa©), quetiapine (Seroquel©), risperidone (Risperdal©), ziprasidone (Geodon©), aripiprazole (Abilify©), asenapine (Saphris©), iloperidone (Fanapt©), lurasidone (Latuda©), haloperidol, chlorpromazine, perphenazine, fluphenazine, thiothixene, or clozapine
* Subjects on other psychoactive medications are asked not to change dose of those medications during the course of the study unless clinically necessary
* Sexually active girls must agree to use two effective forms of birth control (i.e. hormonal or spermicidal and barrier) or be abstinent)
* Primary caretaker is able to participate in study appointments as is clinically indicated
* Ability of child to participate in all aspects of the protocol per investigator's clinical judgment
* After considering all aspects of study participation the subject (if an adult) or subject's parent or Legally Authorized Representative (LAR) must consent to participation
* After considering all aspects of study participation, the subject must assent to participation if it is developmentally appropriate to obtain assent

Exclusion Criteria:

* Based on current or lifetime DSM-IV-TR criteria, a diagnosis of Eating Disorder (Anorexia Nervosa or Bulimia Nervosa)
* Based on DSM-IV-TR criteria, a diagnosis of Substance Dependence Disorder (other than tobacco dependence) within the past month
* Treatment with the following concomitant medications: strong CYP3A4 inhibitors (ex: Ketoconazole), strong CYP3A4 inducers (ex: Rifampin)
* Current or past treatment with lurasidone (Latuda©) that resulted in a non-response or intolerance
* Females who are pregnant or breast-feeding
* Ongoing or previously undisclosed child abuse requiring new department of social service intervention
* Subjects who, in the Investigator's opinion, might not be suitable for the study

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flexible Dose Latuda©
Started | 9
Completed | 7
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Flexible Dose Latuda©
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Change in weight from Baseline to Week 12 will be assessed as the primary outcome measure. Subjects will be asked to step on a special scale called a tanita which will calculate weight, fat mass at each study visit.
Time Frame: Baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: lbs
Arm/Group | Flexible Dose Latuda©
Number analyzed (Participants) | 9
lbs | 0.70 [-5.29 to 6.69]

2. Secondary Outcome: Proportion of Participants Completing Treatment
Description: Data will be collected on why participants terminated the study. If terminated early, the specific reason will be collected such as efficacy or tolerability.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Flexible Dose Latuda©
Number analyzed (Participants) | 9
Participants | 7

3. Secondary Outcome: Changes in Efficacy Measures
Description: Efficacy measures included the Aberrant Behavior Checklist-Community (ABC-C) total score which focuses on problem behaviors in five subdomains, including irritability, attention, repetitive behaviors, unusual speech, and social withdrawal. Differences in subdomains were not assessed. The ABC-C total score is the sum of 58 items, each rated among 0 = Not at all; 1 = Slight in degree; 2 = Moderately serious; and 3 = Severe in degree. The ABC-C total score ranges from 0 to 174. Higher values of ABC-C total scores represent greater severity of illness.
Time Frame: Baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Flexible Dose Latuda©
Number analyzed (Participants) | 9
units on a scale | -14 [-42.76 to 14.76]

4. Secondary Outcome: Number of Participants Experiencing Side Effects
Description: Assessment of the medication side effects associated with lurasidone (Latuda©) in children and adolescents.
Time Frame: Baseline to12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Flexible Dose Latuda©
Number analyzed (Participants) | 9
Participants | 3

5. Secondary Outcome: Overall Clinical Improvement
Description: Overall psychiatric functioning will be assessed with the improvement (CGI-I) subscales of the CGI. CGI-I items are rated from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flexible Dose Latuda©
Number analyzed (Participants) | 9
units on a scale | 2.67 (1.32)

ADVERSE EVENTS:
Arm/Group | Flexible Dose Latuda©
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flexible Dose Latuda© (N=9)
Nausea (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No